CLINICAL TRIAL: NCT01104857
Title: Respiratory Muscle Dysfunction in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Leo Heunks, MD, University Medical Center Nijmegen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Diam1
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Sepsis; Mechanical Ventilation
Keywords: Respiratory muscle; Myosin; Mechanical ventilation
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diaphragm muscle biopsy (Experimental): Patients admitted to the ICU meeting severe sepsis / septic shock criteria
  Interventions: Procedure: diaphragm muscle biopsy
- Elective laparotomy (Active Comparator)
  Interventions: Procedure: Diaphragm muscle biopsy

INTERVENTIONS:
Procedure: diaphragm muscle biopsy — Biopsy is obtained for biochemical analysis
  Arms: Diaphragm muscle biopsy
Procedure: Diaphragm muscle biopsy — Biopsy is obtained for biochemical analysis
  Arms: Elective laparotomy

SUMMARY:
Respiratory muscle dysfunction in critically ill patients is associated with elevated morbidity, including prolonged weaning from mechanical ventilation. The causes for respiratory muscle dysfunction in these patients is poorly understood and no effective treatment is available.

The general hypothesis of the present study is that in critically ill mechanically ventilated subjects respiratory muscle dysfunctions results from loss of myosin induced by activation of proteolytic cascades.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis / septic shock
* Clinical reason for laparotomy
* > 18 years

Exclusion Criteria:

* No informed consent
* Medical history of myopathy
* Unintended weight loss before ICU admission
* Pregnancy
* Chronic use of corticosteroids

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Diaphragm muscle myosin content | 1 day
Markers for inflammation | 1 day
  Inflammatory mediators are measured in plasma and diaphragm at the moment the diaphragm biopsy is obtained.
Markers for activation of proteolytic pathway in the diaphragm | 1 day
  Biochemical analysis is targeted towards activation of several proteolytic pathways (proteasome, lysosmal).

SECONDARY OUTCOMES:
length of ICU stay | 6 months
  Length of ICU stay obtained from medical record
Length of mechanical ventilation | 6 months
  Duration of mechanical ventilation is assesssed within 6 months after obtaining diaphragm biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud Universtity Nijmegen Medical Centre, Nijmegen, Netherlands